CLINICAL TRIAL: NCT05094141
Title: Randomized Pilot Crossover Study Comparing Virtual Reality (VR) and Non-VR Distraction for Decreasing Preoperative/Procedural Anxiety as a Function of the Modified Yale Preoperative Anxiety Scale (mYPAS)
Brief Title: Comparing Virtual Reality (VR) to Non-VR for Decreasing Preoperative/Procedural Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sarah E Rebstock, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STU-2020-0607
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Preoperative Anxiety
Keywords: virtual reality; preoperative anxiety; modified Yale Preoperative Anxiety Scale

STUDY DESIGN:
Intervention Model Description: Randomized Crossover design study will be performed. Subjects will be randomized (1 to 1 randomization) at their initial encounter to either VR or Non-VR. During their second visit patients will be given the alternative mode of care (i.e. patients who initially received VR distraction will be given Non-VR distraction, and patients who initially received Non- VR distraction will receive VR distraction)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-VR (Virtual reality) (No Intervention): The patient is not assigned to play the VR game. mYPAS scoring for port access is done.
- VR (Virtual Reality) (Experimental): The patient is assigned to play the VR game for 15 minutes prior to actual port access procedure start. mYPAS scoring while playing VR device for Port access
  Interventions: Other: Virtual reality

INTERVENTIONS:
Other: Virtual reality — Virtual reality game played during port needle access.
  Other Names: Kind VR game
  Arms: VR (Virtual Reality)

SUMMARY:
The primary objective of the study is to utilize the modified Yale Preoperative Anxiety scale (mYPAS), a validated preoperative/procedural anxiety score, to measure preoperative anxiety via distraction in pediatric oncology patients undergoing port access.

The hypothesis is that using Virtual Reality (VR) will objectively decrease anxiety scores measured by mYPAS by five percent (primary outcome).

The secondary outcome will be the parents or the legally authorized representative (LAR) subjective reports of anxiety with the use of VR.

The Kind VR device is used in house at Children's Health in the Dallas and Plano campuses. The VR device used in this study qualifies as exempt from FDA IDE regulations. It is a non-significant risk, non-invasive, interactive video device the user wears like goggles. The study carries minimal risks to the subjects and is designed to minimize patient discomfort from placement or motion sickness. Furthermore, the device has disposable covers for protection against infection and can be sanitized between uses, once the disposable covers are removed. Children's Health System of Texas (CHST) and this research group are not partnering entities with the Kind VR, and the Kind VR device is not being studied. The effect of virtual reality (VR) on preprocedural anxiety as measured by questionnaires and the observations of the modified Yale Preoperative Anxiety Scale (mYPAS) is being studied

Most patients coming to the Clinic of Cancer and Blood Disorders (CCBD) are under chronic care for their ongoing disease and are likely to be coming to the CCBD at least twice in a 6-month period. The CCBD schedule will be reviewed by the researchers for patients age 5-12, requiring port access at least twice during the next six-month period. Patient families whose child meets the basic screening criteria, and have no exclusion criteria, will be approached privately as possible participants in the study. Up to 100 subjects will be enrolled over a 2-year period. Once the subject/parent or LAR agrees to participate, study staff will randomize the subjects into which standard of care distraction method for anxiety management they will receive first in this study.

DETAILED DESCRIPTION:
1. After the potential participants signed informed consent and were screened for the ability to participate in the study at a treatment appointment.
2. They then came to their cancer center (CCBD) appointment for port access for chemotherapy and were randomized to the Virtual Reality (VR) distraction group first, OR the Non-Virtual Reality (Non-VR) Distraction group first.
3. At this CCBD visit, they then participated in their port needle access as part of standard of care for their cancer treatment using either VR or non-VR distraction for anxiety mitigation, depending on randomization, and were observed during the needle access with the Modified Yale Pre-procedural Anxiety Scale (mYPAS) to assess anxiety during the needle access procedure. The mYPAS is an objective, validated, observational anxiety assessment tool.
4. In addition, parents were asked subjective questions as to how they thought their child tolerated Port needle access with the VR versus Non-VR accordingly.
5. The study personnel then asked when their next potential cancer center appointment for port access to schedule participation in the second arm according to their randomization stratification. In this way, each study participant served as their own control.
6. At the next possible port needle access appointment, they were once again observed using the mYPAS scale for the 2nd port access, with either VR or Non-VR distraction, depending on initial randomization group.
7. Parents were once again asked subjective questions as to how they thought their child tolerated Port needle access with the VR versus Non-VR accordingly.
8. The participants data could Only be included in the study if they participated in both study arms to completion.

ELIGIBILITY:
Inclusion Criteria:

* Any patient of the Children's Medical Center CCBD
* 5-12 years of age
* Patient requiring their port accessed twice or more within a 6 months period
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

* Subjects younger than 5 and older than 12
* Patients requiring recovery in PICU or sites other than PACU
* If parents or subject is not willing to participate
* Subjects with severe developmental delays and subjects with developmental challenges preventing them from keeping the VR device on are also excluded
* Patients who will not be in CCBD for port access at least twice in 6 months

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rebstock, MD, Principal Investigator — UT Southwestern; Neethu Chandran, Principal Investigator — UT Southwestern
Locations (1):
- Kiley Poppino, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fronk E, Billick SB. Pre-operative Anxiety in Pediatric Surgery Patients: Multiple Case Study Analysis with Literature Review. Psychiatr Q. 2020 Dec;91(4):1439-1451. doi: 10.1007/s11126-020-09780-z. PMID 32424544
- [Background] Kain ZN, Mayes LC, Caldwell-Andrews AA, Karas DE, McClain BC. Preoperative anxiety, postoperative pain, and behavioral recovery in young children undergoing surgery. Pediatrics. 2006 Aug;118(2):651-8. doi: 10.1542/peds.2005-2920. PMID 16882820
- [Background] Myers RM, Balsamo L, Lu X, Devidas M, Hunger SP, Carroll WL, Winick NJ, Maloney KW, Kadan-Lottick NS. A prospective study of anxiety, depression, and behavioral changes in the first year after a diagnosis of childhood acute lymphoblastic leukemia: a report from the Children's Oncology Group. Cancer. 2014 May 1;120(9):1417-25. doi: 10.1002/cncr.28578. Epub 2014 Jan 28. PMID 24473774
- [Background] Pelcovitz D, Libov BG, Mandel F, Kaplan S, Weinblatt M, Septimus A. Posttraumatic stress disorder and family functioning in adolescent cancer. J Trauma Stress. 1998 Apr;11(2):205-21. doi: 10.1023/A:1024442802113. PMID 9565912
- [Background] Wu Y, Chen J, Ma W, Guo L, Feng H. Virtual reality in preoperative preparation of children undergoing general anesthesia: a randomized controlled study. Anaesthesiologie. 2022 Dec;71(Suppl 2):204-211. doi: 10.1007/s00101-022-01177-w. Epub 2022 Aug 1. PMID 35925196
- [Background] Agbayani CG, Fortier MA, Kain ZN. Non-pharmacological methods of reducing perioperative anxiety in children. BJA Educ. 2020 Dec;20(12):424-430. doi: 10.1016/j.bjae.2020.08.003. Epub 2020 Oct 21. No abstract available. PMID 33456927
- [Background] Chiu PL, Li H, Yap KY, Lam KC, Yip PR, Wong CL. Virtual Reality-Based Intervention to Reduce Preoperative Anxiety in Adults Undergoing Elective Surgery: A Randomized Clinical Trial. JAMA Netw Open. 2023 Oct 2;6(10):e2340588. doi: 10.1001/jamanetworkopen.2023.40588. PMID 37906193
- [Background] Xu H, Hou J, Zhou J, Wang S. Effects of Virtual Reality on Preoperative Anxiety in Adult Patients: An Updated Meta-analysis. J Perianesth Nurs. 2025 Apr;40(2):422-430.e3. doi: 10.1016/j.jopan.2024.05.009. Epub 2024 Sep 26. PMID 39340515
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Mai CL, Burns S, August DA, Bhattacharya ST, Mueller A, Houle TT, Anderson TA, Peck J. Cardiac index as a surrogate marker for anxiety in pediatric patients undergoing ambulatory endoscopy: a prospective cohort study. Physiol Meas. 2024 Oct 9;45(10). doi: 10.1088/1361-6579/ad805e. PMID 39326507
- [Background] Hu L, Hua Y, Wang L, Mao Z, Jia X, Lei Z, Chang D, Cheng W. Effect of Short-term Deep Breathing Exercises on Perioperative Anxiety and Pain in Pediatric Orthopedic Patients: A Randomized Controlled Trial. J Perianesth Nurs. 2025 Feb;40(1):69-75. doi: 10.1016/j.jopan.2024.03.009. Epub 2024 Jul 9. PMID 38980240
- [Background] Thung A, Tumin D, Uffman JC, Tobias JD, Buskirk T, Garrett W, Karczewski A, Saadat H. The Utility of the Modified Yale Preoperative Anxiety Scale for Predicting Success in Pediatric Patients Undergoing MRI Without the Use of Anesthesia. J Am Coll Radiol. 2018 Sep;15(9):1232-1237. doi: 10.1016/j.jacr.2017.12.022. Epub 2018 Mar 2. PMID 29483054
- [Background] Desai B, Newcomb N, Plost B, Waldron S, Sarkar K, Haber L. Virtual reality use in pediatric patients for orthopedic clinical procedures: A randomized prospective trial of efficacy. J Child Orthop. 2024 May 26;18(4):414-420. doi: 10.1177/18632521241254707. eCollection 2024 Aug. PMID 39100983
- [Background] Chan EA, Chung JW, Wong TK, Lien AS, Yang JY. Application of a virtual reality prototype for pain relief of pediatric burn in Taiwan. J Clin Nurs. 2007 Apr;16(4):786-93. doi: 10.1111/j.1365-2702.2006.01719.x. PMID 17402961
- [Background] Smith KL, Wang Y, Colloca L. Impact of Virtual Reality Technology on Pain and Anxiety in Pediatric Burn Patients: A Systematic Review and Meta-Analysis. Front Virtual Real. 2022 Jan;2:751735. doi: 10.3389/frvir.2021.751735. Epub 2022 Jan 6. PMID 36247202
- [Background] Rodriguez S, Caruso TJ. What every anesthesiologist should know about virtual reality. Paediatr Anaesth. 2022 Dec;32(12):1276-1277. doi: 10.1111/pan.14464. No abstract available. PMID 36352521
- [Background] Tas FQ, van Eijk CAM, Staals LM, Legerstee JS, Dierckx B. Virtual reality in pediatrics, effects on pain and anxiety: A systematic review and meta-analysis update. Paediatr Anaesth. 2022 Dec;32(12):1292-1304. doi: 10.1111/pan.14546. Epub 2022 Sep 1. PMID 35993398

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of patients who were initially enrolled in this randomized crossover design, those not randomized or didn't participate in randomization are reported in the Non-Randomized Arm in the table below.
Groups:
- Non-VR (Virtual Reality), Then VR: The patient is initially assigned to the non-VR group. The non-VR group was the control group defined as the standard of care involving Child Life Guided distractions but not including VR. For both the VR group and the non-VR group, a member of the study team evaluated patient anxiety (using mYPAS) before and during port access--known as the Holding and Induction phases, respectively.
  After the patient completed the first arm of the study (VR or non-VR), the patient was followed for another port access opportunity to complete the alternative study arm depending on initial randomization.
- VR (Virtual Reality), Then Non-VR: The patient is initially assigned to the VR group. The VR group was allowed play the VR game for up to 15 minutes before the port access procedure began and continued to play the game throughout the port access procedure. For both the VR group and the non-VR group, a member of the study team evaluated patient anxiety (using mYPAS) before and during port access--known as the Holding and Induction phases, respectively.
  After the patient completed the first arm of the study (VR or non-VR), the patient was followed for another port access opportunity to complete the alternative study arm depending on initial randomization.
  Virtual reality: Virtual reality game
- Non-Randomized Arm: These patients were enrolled in the study, and had signed an informed consent, but were not randomized.
Period: Overall Study
Arm/Group | Non-VR (Virtual Reality), Then VR | VR (Virtual Reality), Then Non-VR | Non-Randomized Arm
Started | 26 | 26 | 37 (This was a randomized controlled crossover study design. The adverse event - death, due to natural progression of disease in a study participant that was enrolled, had a signed consent, but was NOT randomized.)
Completed | 26 | 26 | 0
Not Completed | 0 | 0 | 37
Not completed — Death | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Subject did not want to wear the VR Helmet | 0 | 0 | 2
Not completed — Did not participate in randomization | 0 | 0 | 33

BASELINE CHARACTERISTICS:
Groups:
- Non-VR (Virtual Reality), Then VR: The patient is not assigned to play the VR game. mYPAS scoring for port access is done.
- VR (Virtual Reality), Then Non-VR: The patient is assigned to play the VR game for 15 minutes prior to actual port access procedure start. mYPAS scoring while playing VR device for Port access
  Virtual reality: Virtual reality game
- Non-Randomized Patients: This group was consented but not randomized into the study.
- Total: Total of all reporting groups
Arm/Group | Non-VR (Virtual Reality), Then VR | VR (Virtual Reality), Then Non-VR | Non-Randomized Patients | Total
Number analyzed (Participants) | 26 | 26 | 37 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 26 | 37 | 89
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 23 | 39
  Male | 18 | 18 | 14 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 5 | 6 | 15
  White | 20 | 19 | 27 | 66
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3
Number of Times of Previous Port Access Procedures [Count of Participants; unit: Participants]
  >10 Times | 15 | 17 | 0 | 32
  7-9 Times | 3 | 1 | 0 | 4
  4-6 Times | 0 | 1 | 0 | 1
  1-3 Times | 4 | 2 | 0 | 6
  0 Times | 4 | 4 | 0 | 8
  Unknown or Not Reported | 0 | 1 | 37 | 38
Taking Medications for Anxiety, Depression, or Agitation [Count of Participants; unit: Participants]
  Yes | 5 | 7 | 0 | 12
  No | 20 | 19 | 0 | 39
  Unknown or Not Reported | 1 | 0 | 37 | 38
History of Claustrophobia [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 0 | 4
  No | 23 | 25 | 37 | 85
History of Motion Sickness [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 0 | 6
  No | 22 | 24 | 37 | 83
Diagnosed with Developmental Delay [Count of Participants; unit: Participants]
  Yes | 2 | 1 | 0 | 3
  No | 24 | 25 | 37 | 86
Likes Playing Video Games [Count of Participants; unit: Participants]
  Yes | 26 | 26 | 0 | 52
  No | 0 | 0 | 37 | 37

OUTCOME MEASURES:

1. Primary Outcome: Preoperative Anxiety Score in Pediatric Oncology Patients
Description: Preoperative anxiety score in pediatric oncology patients as measured by modified Yale Preoperative Anxiety Scale (mYPAS), a validated preoperative/procedural anxiety score.
  Possible scores range from 23 to 100. Higher score values are correlated with increased preoperative anxiety.
Time Frame: 2 years
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- VR (Virtual Reality): The patient is assigned to play the VR game for 15 minutes prior to actual port access procedure start. mYPAS scoring while playing VR device for Port access
  Virtual reality: Virtual reality game
Arm/Group | Non-VR (Virtual Reality) | VR (Virtual Reality)
Number analyzed (Participants) | 52 | 52
score on a scale
  Holding Phase | 31.44 [28.27 to 34.60] | 28.26 [25.81 to 30.71]
  Induction Phase | 45.38 [39.59 to 51.16] | 32.81 [27.88 to 37.74]
  Change from Holding to Induction | 13.94 [8.69 to 19.18] | 4.55 [-0.46 to 9.56]

2. Secondary Outcome: Number of Parents or Legally Authorized Representative (LAR) Who Subjectively Report Decreased Anxiety With the Use of VR
Description: Number of parents or legally authorized representative (LAR) who subjectively report decreased anxiety in their kids (participants in this study) with the use of VR (Virtual Reality) would be calculated based on Parents' questionnaires scored and evaluated for subjective improvement in parental assessment of preoperative anxiety.
Time Frame: 2 years
Population: 51 parents completed the VR experience survey, while one parent opted out of completing the survey. (Only data from parents who completed the VR experience survey have been analyzed and reported for this outcome)
Measure: Number; unit: participants
Arm/Group | Non-VR (Virtual Reality) | VR (Virtual Reality)
Number analyzed (Participants) | 51 | 51
participants
  Holding Phase : Parents Reporting VR Improved Anxiety | 36 | 36
  Holding Phase : Parents Reporting VR Did Not Change Anxiety | 15 | 15
  Holding Phase : Parents Reporting VR Worsened Anxiety | 0 | 0
  Induction Phase : Parents Reporting VR Improved Anxiety | 47 | 47
  Induction Phase : Parents Reporting VR Did Not Change Anxiety | 4 | 4
  Induction Phase : Parents Reporting VR Worsened Anxiety | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Non-ranomized Group: Consented, but never randomized or part of study procedures due to loss to follow up
Arm/Group | Non-VR (Virtual Reality) | VR (Virtual Reality) | Non-ranomized Group
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/52 | 1/37
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/52 | 1/37
Other Adverse Events (participants affected / at risk) | 3/52 | 2/52 | 0/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Non-VR (Virtual Reality) (N=52) | VR (Virtual Reality) (N=52) | Non-ranomized Group (N=37)
mortality (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) — One subject in the Non-randomized group passed away of natural progression of disease after informed consent, but prior to randomization.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-VR (Virtual Reality) (N=52) | VR (Virtual Reality) (N=52) | Non-ranomized Group (N=37)
Dizziness (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 0
Mild headache (General disorders) | 1 | 0 | 0
Nausea (General disorders) | 1 | 0 | 0
Mild rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT05094141/Prot_SAP_000.pdf